CLINICAL TRIAL: NCT04811365
Title: Study Evaluating the Prevalence of the KIT D816V Mutation in Peripheral Blood of Patients With Evidence of Systemic Mast Cell Activation (MCA)
Brief Title: (PROSPECTOR) Screening Study Evaluating the Prevalence of the KIT D816V Mutation in Patients With Systemic Mast Cell Activation
Status: Completed | Type: Observational
Sponsor: Blueprint Medicines Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: BLU-SM-1101
Record Dates: First submitted 2021-03-10; First posted 2021-03-23 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Systemic Mast Cell Activation; KIT D816V Mutation
MeSH Terms: interventions — Mass Screening

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Screening — After providing informed consent, relevant medical history data, and blood and buccal swab samples will be collected at a single visit from patients presenting with systemic mast cell activation symptoms

SUMMARY:
This is a multi-center screening study with the primary objective to determine the prevalence of KIT D816V mutation in peripheral blood in patients with evidence of systemic mast cell activation (MCA).

ELIGIBILITY:
Inclusion Criteria:

* Presenting with at least one of the three criteria below as evidence of systemic mast cell activation:

  1. Involvement of 2 or more organ systems, characterized by skin (pruritus, urticaria, flushing and angioedema), cardiovascular (tachycardia, syncope, and hypotension), gastrointestinal (diarrhea, nausea, vomiting, and gastrointestinal cramping) or respiratory/naso-ocular (wheezing, conjunctival injection, and nasal stuffiness) AND serum basal tryptase levels ≥8 ng/ml. One of the organ systems must be the cardiovascular system.
  2. Severe anaphylaxis (Ring and Messmer grading ≥II) due to Hymenoptera sting, regardless of serum basal tryptase levels.
  3. Severe anaphylaxis (Ring and Messmer grading ≥II), with cardiovascular involvement and documented event-related tryptase elevation fitting the formula 20% of baseline plus 2 ng/ml evaluated in at least 1 event.

Exclusion Criteria:

* Patient previously diagnosed with any of the following WHO systemic mastocytosis (SM) sub-classifications: mastocytosis in the skin, indolent SM, smoldering SM, SM with associated hematological neoplasm, aggressive SM, mast cell leukemia, mast cell sarcoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with systemic mast cell activation
Sampling Method: Non-Probability Sample
Enrollment: 379 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with KIT D816V mutation in peripheral blood | Day 1

SECONDARY OUTCOMES:
Mean KIT D816V mutated allele fraction in peripheral blood | Day 1
Proportion of patients with increased tryptase Alpha/ Beta 1 (TPSAB1) alpha-tryptase gene copy number (GCN) in buccal mucosa | Day 1

CONTACTS AND LOCATIONS:
Locations (23):
- United States (10):
  - Clinical Research Center of Alabama, Birmingham, Alabama
  - Scripps Clinic Carmel Valley, San Diego, California
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Roswell Park Cancer Center, Buffalo, New York
  - Albert P. Hirdt D.O. P.C., New Paltz, New York
  - Columbia University Medical Center - Herbert Irving Comprehensive Cancer Center HICCC, New York, New York
  - Duke University: Duke Allergy Asthma Airway Center, Durham, North Carolina
  - Bernstein Clinical Research Center, LLC, Cincinnati, Ohio
- Antwerp University Hospital UZA, Edegem, Belgium
- France (2):
  - Pitié-Salpêtrière Hospital, Paris
  - CHU Toulouse, Toulouse
- Germany (3):
  - Charite Universitatsmedizin Berlin, Berlin
  - Medizinische Hochschule Hannover, Dept. of Dermatology and Allergy, Hanover
  - Klinik fuer Dermatologie und Allergologie, München
- Italy (2):
  - AOU San Giovanni di Dio e Ruggi d'Aragona University of Salerno, Salerno
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Hospital Virgen del Valle, Toledo, Spain
- University of Basel, Basel, Switzerland
- United Kingdom (3):
  - University Hospital of Leicester, Leicester
  - Guy's and St Thomas' NHS Foundation Trust, London
  - University Hospitals Plymouth NHS Trust, Plymouth